CLINICAL TRIAL: NCT04175288
Title: The Effectiveness of Ultrasound Treatment in the Management of Plantar Fasciitis: A Randomized, Placebo-Controlled Study
Brief Title: The Effectiveness of Ultrasound Treatment in the Management of Plantar Fasciitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Sage Colleges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 802-2019-2020
Record Dates: First submitted 2019-11-15; First posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Plantar Fascitis
MeSH Terms: interventions — High-Energy Shock Waves; Musculoskeletal Manipulations; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound, manual therapy and exercise (Experimental): This group will receive Ultrasound, manual therapy and exercise
  Interventions: Other: Ultrasound, manual therapy and exercise
- manual therapy and exercise (Active Comparator): This group will receive manual therapy and exercise
  Interventions: Other: Ultrasound, manual therapy and exercise

INTERVENTIONS:
Other: Ultrasound, manual therapy and exercise — The experimental group will receive ultrasound (US) for 3 sessions a week for 4 weeks, with continuous US (1.8 w/cm2, 1 Mega Hz 8 minutes). Manual therapy will include posterior glides to talocrural joint, subtalar lateral glide, a 1st tarsometatarsal joint dorsal glide and extension mobilization to the 1st metatarsophalangeal joint. All participants in each group will be given specific exercises by the investgators targeting intrinsic and extrinsic muscles of the foot and ankle. Specific stretches for the plantar fascia and Achilles tendon, will be performed. Home exercises will be recorded using a log.

SUMMARY:
The purpose of this study is to examine the effectiveness of ultrasound treatment in addition to a program consisting of manual therapy and exercise (stretching and strengthening exercises) to improve pain and function in individuals with plantar fasciitis. Our primary hypothesis is individuals with plantar fasciitis will show a greater improvement in pain and function with ultrasound, manual therapy and an exercise program compared to manual therapy and exercise program alone.

DETAILED DESCRIPTION:
Plantar fasciitis (PF) is a common cause of foot pain, affecting an estimated 2 million people per year.1 Although there are large numbers of people seeking medical attention for this condition, there remains some confusion among health care providers as to the most efficacious treatment and some authors conclude that no data solidly supports effectiveness of treatment.2

Several randomized control studies have been published with respect to treatment of PF with ultrasound. The current literature on the effectiveness of US in individuals with PF is largely inconsistent in the parameters. One study by Crawford and Snaith,3 found the true ultrasound was no more effective than sham ultrasound and the authors concluded that future studies need to clarify ultrasound parameters. In contrast, a recent study that utilized different parameters,4 concluded that the US group showed significant changes in pain and function. Strengthening and stretching exercises are well documented through the literature to improve function and decrease pain in patients with PF.5-8 It has been reported within the literature that patients with PF have subtalar, tarsometatarsal, and first metatarsalphangeal (MTP) joint hypo mobility into dorsiflexion, which reduces dorsiflexion range of motion (ROM) and places the windlass mechanism at a mechanical disadvantage which has been theorized to place increased stress on the plantar fascia.9-12 A variety of studies have explored the effects of manual therapy in conjunction with exercises to address the limitations in ankle dorsiflexion ROM.9-12

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above
* onset of plantar heel pain (localized to the medial calcaneal tubercle and have had pain with first steps in the morning)
* both acute and chronic stages of plantar fasciitis

Exclusion Criteria:

* participants currently receiving treatment for plantar fasciitis within the last 6 months including iontophoresis with dexamethasone or acetic acid, corticosteroid injections, extracorporeal shock wave laser therapy, microwave diathermy, radiotherapy, stereotactic radiofrequency, trigger-point needling with infiltration, and ultrasound
* participants that have numbness or tingling with or without provocation in the lower extremity, undiagnosed pain, strength impairment of the ankle of less than a 3+/5 measured with specific manual muscle tests for the gastrocnemius
* participants who are pregnant
* participants who have Type I or II Diabetes Mellitus, systemic inflammatory arthritis, cancer, pacemakers, active tuberculosis, thrombophlebitis, psoriasis, decreased circulation, bleeding disorders or on blood thinning medications, cemented ankle joint replacements, ankle plastic components, acute lower extremity fracture, joint instability and/or hypermobility and osteoporosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11-18 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain during ADL | Change measures (baseline and up to 5 weeks)
  The Numerical Rating Scale/Numerical Pain Rating Scale (NPRS) is a pain scale that has been proven to be a reliable and valid outcome measure when used to assess chronic pain
Range of Motion | Change measures (baseline and up to 5 weeks)
  Dorsiflexion active range of motion will be measured at baseline and at the conclusion of the study by the other principal investigator. Participants will be in a weight-bearing lunge position with the leg to be measured in front and toes facing the wall. The participant will be asked to maximally bend the knee without lift of the heel.
Functional foot and ankle measure (ADL and sports) | Change measures (baseline and up to 5 weeks)
  The Foot and Ankle Ability Measure (FAAM) is a functional outcome measure validated in the physical therapy setting.20 It will be used to measure differences in ability in activities of daily living and sports at the initial evaluation and at the conclusion of the study.
Heel raises | Change measures (baseline and up to 5 weeks)
Navicular drop | Change measures (baseline and up to 5 weeks)
  All subjects will be seated in a chair with the hips and knees flexed to 90 degrees. The subtalar joint neutral position will be 1st identified through appropriate technique. Following this, the examiner will identify the most anterior and inferior position of the navicular tuberosity and mark it with a washable fine tip marker. The participant will be asked to hold that position while the height of the navicular tuberosity will be measured with a digital caliper. Following measurements in seated position for both feet, participants will be asked to stand and assume a relaxed stance position. The process measuring the navicular height position with a digital caliper as described above in seated position will be repeated in standing position. The difference between the seated and standing navicular positions will be defined as the Navicular drop.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Elkins, Principal Investigator — The Sage Colleges
Locations (1):
- Neeti Pathare, Troy, New York, United States

IPD SHARING:
Plan to Share IPD: No